CLINICAL TRIAL: NCT03613688
Title: Effects of Deepure(Pu-erh Tea Extract) on Glycemic Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tasly Pharmaceuticals, Inc. (Industry)
Collaborators: Natural Immune Systems Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 079-007
Record Dates: First submitted 2018-07-26; First posted 2018-08-03 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Glucose Metabolism Disorders
MeSH Terms: conditions — Glucose Metabolism Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Deepure Group A (Experimental): Visit 3: Warm water without Deepure; Visit 4: Warm water with 1 g Deepure; Visit 5: Warm water with 1.5 g Deepure; Visit 6: Warm water with 2 g Deepure.
  Interventions: Dietary Supplement: Deepure
- Deepure Group B (Experimental): Visit 3: Warm water with 1 g Deepure; Visit 4: Warm water with 1.5 g Deepure; Visit 5: Warm water with 2 g Deepure; Visit 6: Warm water without Deepure.
  Interventions: Dietary Supplement: Deepure
- Deepure Group C (Experimental): Visit 3: Warm water with 1.5 g Deepure; Visit 4: Warm water with 2 g Deepure; Visit 5: Warm water without Deepure; Visit 6: Warm water with 1 g Deepure.
  Interventions: Dietary Supplement: Deepure
- Deepure Group D (Experimental): Visit 3: Warm water with 2 g Deepure; Visit 4: Warm water without Deepure; Visit 5: Warm water with 1 g Deepure; Visit 6: Warm water with 1.5 g Deepure.
  Interventions: Dietary Supplement: Deepure

INTERVENTIONS:
Dietary Supplement: Deepure — Pu'erh Tea extract

SUMMARY:
This is a randomized, controlled, cross-over study on the effects of consumption of Deepure puerh tea extract (PTE) on glucose tolerance and metabolic markers.

DETAILED DESCRIPTION:
The study will involve consuming three different doses: 1 gram, 1.5 grams, and 2 grams, and will be given in warm water, with a bland meal. The effects on glucose and insulin after consumption will be evaluated.The subjects will be randomly assigned to one of four groups with different sequences.

ELIGIBILITY:
Inclusion Criteria:

* Men and women;
* Aged 18-70 years;
* BMI between 20-30;
* Fasting blood glucose at screening between 71-125 mg/dL. both inclusive.

Exclusion Criteria:

* Taking dietary supplements judged to interfere with the effects of Deepure on glucose metabolism (for example: cinnamon extract; chromium picolinate; mulberry extract; bitter melon extract, green tea extracts, black tea extracts, pu-erh tea);
* Participation in other clinical trials, involving an investigational product or lifestyle change, during the last month;
* Participation in another research study during this trial, involving an investigational product or lifestyle change; Taking prescription medication known to affect glucose metabolism;
* Taking over-the-counter medication known to affect glucose metabolism;
* Drinking 3 or more cups of tea daily;
* Unwilling to abstain from drinking tea for 24 hours before clinic visits; (if a person drinks tea within 24 hours of a clinic visit, the person's visit will be re-scheduled);
* Consuming 2 or more drinks of alcohol per day;
* Unwilling to abstain from drinking alcohol for 10 hours before clinic visits;
* Diagnosed with diabetes Type I; Taking medication for diabetes Type II;
* Diagnosed with the thyroid disorder Hashimoto's disease;
* Past major surgery to your stomach or intestines (minor surgery not a problem such as hernia repair, appendix removal, gallbladder removal);
* Currently taking cholesterol-lowering medication (for example: statins);
* Currently taking coumadin;
* Major trauma within the past 6 months;
* Major surgery within the past 6 months;
* Severe chronic infectious disease (such as HIV, chronic hepatitis);
* Active depression;
* Self-reported eating disorders;
* History of drug abuse during past two years;
* Currently going through intense stressful events or life changes;
* Women of child-bearing potential: Pregnant, breast-feeding, or trying to become pregnant;
* Women of child-bearing potential: Not using effective contraception;
* Food allergies or sensitivities to tea.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2018-09-20 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Post-prandial glucose response | From baseline to 30, 60, 90, 120, and 180 minutes
  Change in blood glucose leve after consuming test meal with and without Pu'er tea

CONTACTS AND LOCATIONS:
Locations (1):
- NIS labs, Klamath Falls, Oregon, United States

IPD SHARING:
Plan to Share IPD: No